CLINICAL TRIAL: NCT03412344
Title: Assessing Knowledge and Affecting Factors Associated With Cancer Patients Participation in Clinical Trials in China.
Brief Title: Factors Influencing Cancer Patients Participation in Clinical Trials in China.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, Professor of medical oncology Deputy Director National Cancer Center Vice President Cancer Hospital Chinese Academy of Medical Sciences(CAMS) & Peking Union Medical College(PUMC), Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: CH-HUR-004
Record Dates: First submitted 2017-12-29; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Cancer
Keywords: clinical trial; patient; questionnaire
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research studies factors affecting Chinese patient participation in cancer clinical trials and their knowledge regarding clinical trials. The investigators design this study to determining how patients makes decisions about participating in a clinical trial and know about patients' attitude toward clinical trials. The investigators aim to find ways to make cancer clinical trials in China more efficient and satisfied patients participating in clinical trials in China.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of malignancy
* Aged 18 years or older
* Ability to understand and complete the questionnaire independently or with the help of a relative or staff member of the oncology department
* Patients have been consented to join an oncology treatment clinical study and have begun active treatment of an oncology clinical trial

Exclusion Criteria:

• Not meeting all eligibility criteria

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese patients with a diagnosis of cancer who have joined cancer clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The patient related factors and the doctor related factors that influence patient decision regarding participation in a cancer clinical trial will be explored by questionnaire. | 1 year

SECONDARY OUTCOMES:
Oncology patients' understanding and attitude of clinical trials towards cancer clinical research will be evaluated by questionnaire. | 1 year
The actual experience of participants in a cancer clinical trial will be investigated by questionnaire. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, PhD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jiang S, Liu P, Yang S, Yang J, Wu D, Fang H, Qin Y, Zhou S, Xu J, Sun Y, Mo H, Gui L, Xing P, Lan B, Zhang B, Tang L, Sun Y, Shi Y. Evaluating stress, satisfaction and the associated influencing factors of participants in cancer clinical trials: a cross-sectional study in China. BMJ Open. 2019 Jun 1;9(5):e028589. doi: 10.1136/bmjopen-2018-028589. PMID 31154312